CLINICAL TRIAL: NCT05223647
Title: Randomized Phase III Trial Investigating the Survival Benefit of Adding Thoracic Radiotherapy to Durvalumab (MEDI4736) Immunotherapy Plus Chemotherapy in Extensive Stage Small-cell Lung Cancer
Brief Title: Chemo-immunotherapy Plus Thoracic Radiotherapy in Extensive Stage Small-cell Lung Cancer
Acronym: TRIPLEX
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Termination was adviced by Data Safety Committee due to excess toxicity of the experimental treatment.
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); Haukeland University Hospital (Other); University Hospital of North Norway (Other); Alesund Hospital (Other); Helse Stavanger HF (Other Government); Oslo University Hospital (Other); Helse Nord-Trøndelag HF (Other); Helse Fonna (Other); Drammen sykehus (Other); University Hospital, Akershus (Other); Erasmus Medical Center (Other); Sahlgrenska University Hospital (Other); Karolinska University Hospital (Other); Gävle Hospital (Other); Sykehuset Innlandet HF (Other); North Estonia Medical Centre (Other); Nordlandssykehuset HF (Other); Landspitali University Hospital (Other); Lund University Hospital (Other); University Hospital, Linkoeping (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EC#230766; 2020203 (Other Grant/Funding Number: Clinical therapy research in the specialist health services)
Record Dates: First submitted 2022-01-11; First posted 2022-02-04 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Small-cell Lung Cancer
Keywords: cancer; chemotherapy; radiotherapy; immunotherapy
MeSH Terms: conditions — Small Cell Lung Carcinoma; Neoplasms | interventions — Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chemo-immunotherapy plus thoracic radiotherapy (Experimental): Four courses of carboplatin/etoposide/durvalumab every 3 weeks followed by durvalumab every 4 weeks until intolerable toxicity, progressive disease leading to a need for other treatment, or until the patient no longer wishes to continue treatment.
  Thoracic radiotherapy of 30 Gy/10 fractions between 2nd and 3rd carboplatin/etoposide/durvalumab course.
  Interventions: Procedure: Thoracic radiotherapy; Drug: Chemo-immunotherapy
- Chemo-immunotherapy (Active Comparator): Four courses of carboplatin/etoposide/durvalumab every 3 weeks followed by durvalumab every 4 weeks until intolerable toxicity, progressive disease leading to a need for other treatment, or until the patient no longer wishes to continue treatment.
  Interventions: Drug: Chemo-immunotherapy

INTERVENTIONS:
Procedure: Thoracic radiotherapy — 30Gy/10 fractions thoracic radiotherapy given between 2nd and 3rd course of chemo-immunotherapy.
  Arms: Chemo-immunotherapy plus thoracic radiotherapy
Drug: Chemo-immunotherapy — Four courses of carboplatin/etoposide/durvalumab every 3 weeks followed by durvalumab every 4 weeks until intolerable toxicity, progressive disease leading to a need for other treatment, or until the patient no longer wishes to continue treatment.
  Other Names: carboplatin/etoposide/durvalumab

SUMMARY:
Studies have shown that combining chemotherapy and immune checkpoint inhibitors (ICI) prolongs survival compared with chemotherapy alone in extensive stage small-cell lung cancer (ES SCLC), but the survival benefit is modest. The main aim of this trial is to investigate whether there is a synergistic/additive effect of concurrent thoracic radiotherapy in ES SCLC patients receiving carboplatin/etoposide/durvalumab.

DETAILED DESCRIPTION:
Studies show that adding ICI therapy to standard chemotherapy prolongs survival in ES SCLC. The survival benefit, however, is modest, and there is a need for more effective therapy. It has been hypothesized that there is a synergistic effect of combining ICI with radiotherapy. In this randomized phase III study, the main aim is to investigate whether concurrent thoracic radiotherapy of 30 Gy/10 fractions improves survival in ES SCLC patients receiving carboplatin/etoposide/durvalumab.

It is currently not possible to classify the patients who benefit from ICIs in SCLC. In this study, biological material (tissue, blood, feces) which will be analyzed for potential predictive and prognostic biomarkers.

Prophylactic cranial irradiation in ES SCLC is debated, mainly due to the potentially detrimental effect on cognition. Thus, frequency and timing of brain metastases and cognitive function will be assessed before, during and after study treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years at time of study entry
2. ECOG performance status of 0 or 1
3. Body weight >30 kg
4. Adequate bone marrow, liver and kidney function
5. Life expectancy of at least 3 months
6. At least one measurable (RECIST 1.1), thoracic lesion that can be irradiated with 30 Gy/10 fractions
7. Histologically or cytologically confirmed SCLC
8. Stage III-IV disease (TNM v8)
9. FEV1 >1 L or >30 % of predicted value and DLCO >30 % of predicted value
10. Patients with brain metastases are eligible provided they are asymptomatic or treated and stable on steroids and/or anticonvulsants prior to the start of treatment

Exclusion Criteria:

1. Previous chemo-, immuno- or radiotherapy for SCLC
2. Major surgical procedure last 28 days
3. History of allogenic organ transplantation, autoimmune disease, immunodeficiency, hepatitis or HIV
4. Uncontrolled intercurrent illness
5. Other active malignancy
6. Leptomeningeal carcinomatosis
7. Immunosuppressive medication
8. Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2022-01-11 (Actual); Primary Completion 2025-09-04 (Actual); Study Completion 2025-09-04 (Actual)

PRIMARY OUTCOMES:
Change in 1-year overall survival | 14 months after last patient entry
  The Cox proportional hazards method will be used to compare survival between the treatment groups.

SECONDARY OUTCOMES:
Change in 2-, 3-, 4- and 5-year survival rate | 2, 3, 4 and 5 years after last patient entry
  The Cox proportional hazards method will be used to compare survival between the treatment groups.
Frequency and severity of adverse events | Through study completion, an average of 1 year after last patient entry
  Adverse events will be compared between the treatment arms using the Pearson's Chi-square and Fisher's exact test.
Change in progression free survival (PFS) | Through study completion, an average of 1 year after last patient entry
  PFS will be estimated using the Kaplan-Meier method and compared using the log-rank test. A Cox-model adjusting for baseline characteristics will be used for multivariable analyses.
Change in overall response rates | Through study completion, an average of 1 year after last patient entry
  Response rates are compared using Pearson's Chi-square test.
Change in response rates in non-irradiated lesions | Through study completion, an average of 1 year after last patient entry
  Response rates are compared using Pearson's Chi-square test.
Local control rates in the thorax | Through study completion, an average of 1 year after last patient entry
  Local control rates are compared using Pearson's Chi-square test.
Health-related quality of life (HRQoL) | Through study completion, an average of 1 year after last patient entry
  All HRQoL scores will be transformed to a scale of 0-100 according to the EORTC QLQ scoring manual. Mean scores will be compared at each assessment timepoint, and a difference of 10 points is considered clinically relevant.

OTHER OUTCOMES:
Change in cognitive function from baseline to end of treatment | Through study completion, an average of 2 years after last patient entry
  Cognitive function will be compared between patients who receive PCI and those who do not, using the MoCA-test. Scores will be compared using the Mann-Whitney test.
Frequency and timing of brain metastases | Through study completion, an average of 2 years after last patient entry
  Changes in brain metastases are compared using Pearson's Chi-square test.
Associations between outcomes of study treatment and biomarkers in tissue, blood and stool | Through study completion, an average of 2 years after last patient entry
  A detailed plan for analyses will be defined when sufficient material for translational research has been collected.

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Steigedal, PhD, Study Director — Department of Clinical and Molecular Medicine, NTNU
Locations (20):
- North Estonia Medical Centre, Tallinn, Estonia
- Landspitali University Hospital, Reykjavik, Iceland
- Erasmus MC, Rotterdam, Netherlands
- Norway (12):
  - Ålesund Hospital, Ålesund
  - Haukeland Universitetssykehus, Bergen
  - Nordlandssykehuset HF, Bodø
  - Drammen sykehus - Vestre Viken, Drammen
  - Innlandet hospital Gjøvik, Gjøvik
  - Haugesund hospital, Haugesund
  - Sykehuset Levanger, Levanger
  - Akershus Universitetssykehus AHUS, Oslo
  - Oslo University Hospital Ullevål, Oslo
  - Stavanger University Hospital, Stavanger
  - University Hospital of North Norway, Pulmonology Department, Tromsø
  - Cancer Clinic at St. Olavs Hospital, Trondheim
- Sweden (5):
  - Gävle hospital, Gävle
  - Sahlgrenska Sjukehuset, Gothenburg
  - Linköping University Hospital, Linköping
  - Lund University Hospital, Skåne
  - Karolinska University Hospital, Stockholm

IPD SHARING:
Plan to Share IPD: Yes
Results, including biomarker analyses, will be made available in Sponsor's data repository based on the data management plan and according to FAIR principles.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: December 2029
Access Criteria: The repository is based on Dataverse, and available for anyone.

DOCUMENTS (2):
  • Study Protocol (2022-01-05): https://cdn.clinicaltrials.gov/large-docs/47/NCT05223647/Prot_000.pdf
  • Informed Consent Form (2021-12-21): https://cdn.clinicaltrials.gov/large-docs/47/NCT05223647/ICF_001.pdf